CLINICAL TRIAL: NCT02201264
Title: The Atlantic CPORT Primary PCI Registry
Brief Title: Cardiovascular Patient Outcomes and Research Team Primary PCI Registry
Acronym: CPORT
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 11.2
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: myocardial infarction; Angioplasty; Stent
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary PCI for STEMI patients: Primary PCI for patients presenting with ST elevation MIs

SUMMARY:
The proposed study is a registry of patients treated with primary angioplasty for acute myocardial infarction.

The aim of this registry is to define the outcomes of patients treated for acute, ST-segment myocardial infarction (STEMI) at community hospitals without on-site cardiac surgery programs that have completed the Cardiovascular Patient Outcomes and Research Team (C-PORT) Primary Angioplasty Development program. The primary medical outcome for the registry is the combined incidence of death, recurrent non-fatal myocardial infarction and stroke.

DETAILED DESCRIPTION:
The primary study endpoint is the composite incidence of death, non-fatal reinfarction and stroke 6 weeks after index myocardial infarction.

Secondary endpoints include:

1. composite of death, recurrent non-fatal MI and stroke at hospital discharge and at 6 months
2. specific subgroup analyses are planned based on history of diabetes age anterior versus other infarct locations race gender
3. incidence of complications including significant bleeding, need for coronary artery bypass surgery, cardiac arrest

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years
2. ability to give informed consent
3. acute myocardial infarction with

   1. > 30 mins ongoing ischemic cardiac pain at presentation and > 0.1 mv ST-segment elevation in 2 or more contiguous ECG leads or
   2. new or suspected new Left Bundle Branch Block (LBBB) or
   3. > 0.1 mv ST-segment depression in V1 and V2 consistent with true posterior infarction
4. rescue PCI for failed thrombolytics
5. cardiogenic shock - (defined as systolic blood pressure <80 mmHg sustained for more than 30 minutes despite correction of non-myocardial factors (hypovolemia, acidosis, arrhythmia, etc) or requirement for pressors and/or intra-aortic balloon pump (IABP) to sustain systolic blood pressure > 80 mmHg)

Exclusion Criteria

1. inability to obtain informed consent (surrogate consent may be obtained if approved by your IRB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute myocardial infarction with
  1. > 30 mins ongoing ischemic cardiac pain at presentation and > 0.1 mv ST-segment elevation in 2 or more contiguous ECG leads or
  2. new or suspected new LBBB or
  3. > 0.1 mv ST-segment depression in V1 and V2 consistent with true posterior infarction cardiogenic shock - (defined as systolic blood pressure <80 mmHg sustained for more than 30 minutes despite correction of non-myocardial factors (hypovolemia, acidosis, arrhythmia, etc) or requirement for pressors and/or IABP to sustain systolic blood pressure > 80 mmHg)
Sampling Method: Non-Probability Sample
Enrollment: 6726 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Composite incidence of death, non-fatal reinfarction and stroke. | 6 weeks after myocardial infarction
  The primary study endpoint is the composite incidence of death, non-fatal reinfarction and stroke 6 weeks after index myocardial infarction.
  Secondary endpoints include:
  1. composite of death, recurrent non-fatal MI and stroke at hospital discharge and at 6 months
  2. specific subgroup analyses are planned based on history of diabetes age anterior versus other infarct locations race gender
  3. incidence of complications including significant bleeding, need for coronary artery bypass surgery, cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aversano, MD, Study Director — Johns Hopkins School of Medicine
Locations (14):
- United States (14):
  - Community Health and Wellness Center, Bryan, Ohio
  - University Hospital Geauga Medical Center, Chardon, Ohio
  - Ohio State University East, Columbus, Ohio
  - Southview Medical Center, Dayton, Ohio
  - Fort Hamilton Hospital, Hamilton, Ohio
  - Marietta Memorial, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Westchester Hospital, Westchester, Ohio
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - UPMC McKeesport, McKeesport, Pennsylvania
  - Meadville Medical Center, Meadville, Pennsylvania
  - Nazareth Hospital, Philadelphia, Pennsylvania
  - Memorial Hospital, York, Pennsylvania